CLINICAL TRIAL: NCT01633749
Title: Immunogenicity, Reactogenicity and Safety of the Trivalent Influenza Subunit Vaccine Influvac® for the Northern Hemisphere Season 2012/2013. An Open-label, Baseline-controlled Study in Two Age Groups: Adult Subjects ≥ 18 and ≤ 60 Years and Elderly Subjects ≥ 61 Years of Age
Brief Title: Annual Study to Investigate Inactivated Subunit Influenza Vaccine Due to New Virus Strains for the 2012/2013 Season
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Biologicals (Industry)
Responsible Party: Sponsor
Organization: Abbott (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: M13-567; 2012-001032-57 (EudraCT Number)
Record Dates: First submitted 2012-07-02; First posted 2012-07-04 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Prophylaxis of Influenza
Keywords: Influenza; Vaccine; CHMP criteria
MeSH Terms: conditions — Influenza, Human | interventions — influvac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trivalent influenza subunit vaccine Influvac (Experimental): 3x 15mcg HA per 0.5 ml,trivalent one injection at Day 1
  Interventions: Biological: Trivalent influenza subunit vaccine Influvac

INTERVENTIONS:
Biological: Trivalent influenza subunit vaccine Influvac — 3x 15mcg HA per 0.5 ml,trivalent one injection at Day 1
  Other Names: ABT-SLV201, trivalent influenza subunit vaccine, Influvac

SUMMARY:
Annual study to investigate influenza vaccine (flu vaccine) developed for the 2012/2013 season for the prevention of influenza infection. The immunizing effect is being investigated, as well as its tolerability and safety.

DETAILED DESCRIPTION:
An open, baseline-controlled study in two age groups: adults and elderly. The subjects will be screened within 14 days prior to or at Visit 1 (Day 1). At Visit 1 (Day 1) subjects will be vaccinated after blood sampling for baseline serum antihemagglutinin antibody titration. Subjects will be asked to record local and systemic reactions daily on a diary at home for 72 hours after vaccination. One week later (Visit 2, Day 8) the subjects will return to the study site to hand in the diary and for the assessment of safety and tolerability (reactogenicity and overall inconvenience). Three weeks after vaccination (Visit 3, Day 22) the subjects will return to the study site for blood sampling to assess immunogenicity and for the assessment of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria

1. Willing and able to give informed consent and able to adhere to all protocol required study procedures.
2. Men and women aged ≥ 18 and ≤ 60 years or ≥ 61 years of age at the day of study vaccination.
3. Being in good health as judged by medical history, physical examination (if needed) and clinical judgment of the Investigator.

Exclusion Criteria

1. Known to be allergic to eggs, chicken protein, gentamicin or any other constituent of the vaccine.
2. A serious adverse reaction after a previous (influenza) vaccination.
3. Presence of any significant condition that may prohibit inclusion as determined by the investigator.
4. Seasonal or pandemic influenza vaccination or laboratory confirmed seasonal or pandemic influenza infection within the previous six months before study vaccination or planned vaccination during the study period.
5. Having any condition which suppresses the immune system and autoimmune disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Antihemagglutinin antibody titers and the derived parameters seroprotection, seroconversion and mean fold increase | 3 weeks
  Standard parameters to quantify antibody levels. Recommended in the CHMP guideline.
Solicited local and systemic reactions, overall inconvenience | 3 days
  Reactogenicity and inconvenience
Unsolicited adverse events | 3 weeks
  Other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Serge van de Witte, PhD, Study Director — Abbott Healthcare Products BV
Locations (1):
- Site Reference ID/Investigator# 74593, Hamburg, Germany